CLINICAL TRIAL: NCT00002544
Title: MITOXANTRONE (N) VS. 5-FLUOROURACIL, EPIRUBICIN AND CYCLOPHOSPHAMIDE AS FIRST-LINE CHEMOTHERAPY FOR PATIENTS WITH METASTATIC BREAST CANCER AND AN UNFAVORABLE PROGNOSIS
Brief Title: Mitoxantrone With or Without Docetaxel in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbeitsgemeinschaft fur Internistische Onkologie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GER-AIO-01/92; CDR0000063279 (Registry Identifier: PDQ (Physician Data Query)); EU-93011
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2001-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Mitoxantrone

INTERVENTIONS:
Drug: docetaxel
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if mitoxantrone is more effective with or without docetaxel.

PURPOSE: Randomized phase III trial to compare the effectiveness of mitoxantrone with or without docetaxel in treating women who have metastatic breast cancer with a poor prognosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival and quality of life scores (composed of time to progression, WHO performance status, subjective patient evaluation, and subjective adverse event profile) among women with metastatic breast cancer of unfavorable prognosis treated with mitoxantrone vs mitoxantrone plus docetaxel as first-line chemotherapy for metastatic disease.
* Compare the remission rate, time to remission, remission duration, time to best response, objective adverse events, and patient acceptance of treatment on these 2 regimens.
* Investigate which prognostic subgroups of women benefit from treatment.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age, treatment center, disease free interval (no more than 18 months vs more than 18 months), hormone receptor status (positive or unknown vs negative), prior adjuvant therapy with anthracyclines (yes vs no), presence of liver metastases (liver involvement as a single organ vs liver plus other organ involvement vs no liver involvement), and presence of lung metastases (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive mitoxantrone IV on day 1. Treatment repeats every 3 weeks until disease progression, unacceptable toxicity, or maximum cumulative dose. Patients who achieve complete response receive 2 additional courses.
* Arm II: Patients receive mitoxantrone IV plus docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

At relapse, reinduction with the original regimen is attempted. Following a second complete response, 2 additional courses of consolidative treatment are given, and patients are then followed off treatment.

Quality of life is assessed periodically.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic breast cancer of poor prognosis, defined by any of the following characteristics:

  * Patient aged 35 or under
  * Liver metastases
  * Lung metastases combined with other disease manifestations
  * Lung metastases without other disease manifestations but with a disease free interval of no more than 18 months
* Indication for chemotherapy documented by either:

  * Hormone receptor negativity OR
  * Hormone resistant disease
* Measurable metastatic disease required

  * Nonmeasurable disease includes:

    * Metastases verified only histologically
    * Tumor parameters not precisely measurable (e.g., bone marrow involvement, lymphangitic disease)
* No CNS metastasis or bone marrow carcinomatosis
* Hormone receptor status:

  * Receptor status known

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC greater than 4,000/mm^3
* Absolute granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 6 times ULN
* SGOT and/or SGPT no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.15 times ULN

Cardiovascular:

* No uncontrolled hypertension
* No congestive heart failure within the past 6 months
* No myocardial infarction within the past 6 months

Other:

* Fertile patients must use effective contraception
* No acute or chronic infection
* No second primary tumor
* No other serious illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy for metastatic disease
* Greater than 1 year since prior adjuvant chemotherapy
* No prior anthracycline or anthraquinone

Endocrine therapy:

* Hormone resistant disease required of receptor positive patients
* No concurrent endocrine therapy

Radiotherapy:

* No prior mediastinal irradiation
* Adjuvant irradiation of parasternal nodes eligible
* No prior irradiation to more than 25% of bone marrow
* No concurrent irradiation of sole measurable lesion

Surgery:

* Not specified

Other:

* No concurrent anticoagulant therapy

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1993-05; Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Else G. Heidemann, MD, Study Chair — Diakonie-Klinikum Stuttgart
Locations (1):
- Diakonissen-Krankenhaus Stuttgart, Stuttgart, Germany

REFERENCES:
- [Background] Heidemann E, Souchon R, Stoger H, et al.: First-line monochemotherapy with mitoxantrone versus combination with fluorouracil, epirubicin and cyclophosphamide in high-risk metastatic breast cancer: a prospective randomized multicenter clinical trial. Onkologie 23(1): 54-59, 2000.
- [Background] Heidemann E, Stoeger H, Souchon R, et al.: Balance of time to progression, quality of life, and overall survival: more gain from treatment in single agent treatment with mitoxantrone (N) than with the combination of fluorouracil, epirubicin, cyclophosphamide (FEC). Results of a multicenter randomized trial in high risk metastatic breast cancer (MBC). [Abstract] Proceedings of the American Society of Clinical Oncology A-284, 74a, 2000.
- [Background] Loibl S, von Minckwitz G, Souchon R, et al.: Phase I/II study with mitoxantrone (N) vs. NDOC in patients with high risk locally advanced or metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A512, 1999.
- [Result] Heidemann E, Stoeger H, Souchon R, Hirschmann WD, Bodenstein H, Oberhoff C, Fischer JT, Schulze M, Clemens M, Andreesen R, Mahlke M, Konig M, Scharl A, Fehnle K, Kaufmann M. Is first-line single-agent mitoxantrone in the treatment of high-risk metastatic breast cancer patients as effective as combination chemotherapy? No difference in survival but higher quality of life were found in a multicenter randomized trial. Ann Oncol. 2002 Nov;13(11):1717-29. doi: 10.1093/annonc/mdf306. PMID 12419743